CLINICAL TRIAL: NCT01379989
Title: Phase III International, Randomized Study of Trabectedin Plus Pegylated Liposomal Doxorubicin (PLD) Versus Carboplatin Plus PLD in Patients With Ovarian Cancer Progressing Within 6-12 Months of Last Platinum
Brief Title: INOVATYON STUDY -International, Randomized Study in Patients With Ovarian Cancer
Acronym: INOVATYON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: PharmaMar (Industry); Averion International Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET-D-009-10
Record Dates: First submitted 2011-06-01; First posted 2011-06-23 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; liposomal doxorubicin; Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin plus PLD (Active Comparator): Pegylated Lipoxomal Doxorubicin (PLD) 30 mg/ m2 followed by carboplatin AUC 5.
  Interventions: Drug: Carboplatin; Drug: Pegylated Lipoxomal Doxorubicin (PLD)
- Trabectedin plus PLD (Experimental): Pegylated Lipoxomal Doxorubicin (PLD) 30 mg/m2 infusion followed by trabectedin 1.1 mg/m2 infusion.
  Interventions: Drug: Pegylated Lipoxomal Doxorubicin (PLD); Drug: Trabectedin

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC 5
  Other Names: Carboplatin generic
  Arms: Carboplatin plus PLD
Drug: Pegylated Lipoxomal Doxorubicin (PLD) — PLD 30 mg/m² i.v.
  Other Names: Caelyx
Drug: Trabectedin — trabectedin 1.1 mg/m2 3-hour i.v. infusion on Day 1 every 3 weeks. The use of central venous access is strongly recommended.
  Other Names: Yondelis
  Arms: Trabectedin plus PLD

SUMMARY:
The objective of this multicentric, randomised, Phase III study is to demonstrate superiority, in terms of survival, of trabectedin and Pegylated Liposomal Doxorubicin (PLD) versus carboplatin and PLD in partially-platinum sensitive ovarian cancer patients.

DETAILED DESCRIPTION:
Patients will be randomised to:

Arm A: PLD 30 mg/m2 and carboplatin AUC 5; Arm B: PLD 30 mg/m2 and trabectedin 1.1 mg/m2. Patients' characteristics: patients over 18 years of age with advanced, progressive ovarian cancer 6-12 months after completion of first line or second line treatment with platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged ≥ 18 years
2. Histologically and/or cytologically proven epithelial ovarian, epithelial fallopian tube cancer or primary peritoneal cancer
3. Progression free interval between six and twelve (6-12) months (calculated from the first day of the last cycle of the last platinum-based chemotherapy until the date of progression confirmation through radiologic imagery). Patients may have received up to two platinum-based chemotherapy lines, of which at least one must have contained a taxane
4. Measurable or evaluable disease confirmed by radiological imaging, such as magnetic resonance imaging (MRI), computed tomography (CT) scan, or PET/CT scan at study entry (CA-125 rise not supported by radiological evidence of disease is not accepted as criteria for defining progression) or histological proven recurrent ovarian cancer even in the absence of postoperatively measurable or evaluable lesions.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
6. Estimated life expectancy ≥ 12 weeks
7. Patients must be accessible for treatment and follow-up
8. Adequate organ function within 14 days prior to first cycle as evidenced
9. Patients must be able to receive dexamethasone or its equivalent, which is required if randomly assigned to treatment with trabectedin plus PLD
10. Informed consent of the patient

Exclusion Criteria:

1. Non epithelial ovarian or mixed epithelial/non epithelial tumors (e.g., Mullerian tumors)
2. Patients who did not respond to last platinum-based therapy or in whom last relapse occurred < 6 months or > 12 months from the last dose of platinum
3. Bowel obstruction, sub-occlusive disease or the presence of symptomatic brain metastases
4. Pre-existing grade > 1 motor or sensory neuropathy according to the National Cancer Institute Common Toxicity Criteria Adverse Event (NCI-CTCAE) version 4.0
5. Myocardial infarct within six months before enrolment, New York Association (NYHA) Class II or worse heart failure (Appendix 1. The New York Heart Association), uncontrolled angina, severe uncontrolled ventricular arrythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
6. History of liver disease
7. Concurrent severe medical problems or any unstable medical condition unrelated to malignancy, which would significantly limit full compliance with the study or expose the patient to extreme risk or decreased life expectancy
8. Breastfeeding women and women of child bearing potential must use effective contraception during treatment and 3 months thereafter, which may include prescription contraceptives (oral, injection, or patch), intrauterine device, double-barrier method or male partner sterilization (not applicable to patients that are surgically sterile)
9. Prior exposure to trabectedin
10. Prior resistance to anthracyclines or PLD defined as a progression during anthracycline-based chemotherapy or a recurrence within 6 months from its ending
11. Prior severe PLD related toxicity
12. Prior exposure to cumulative doses of doxorubicin >400mg/m2 or epirubicin >720mg/m2
13. Treatment with any investigational product within 30 days prior to inclusion in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2011-06; Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled
  This is an event driven study. The study will continue until 442 events have occurred.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  PFS will be measured from the date of randomization to the date of documented PD or death (regardless of cause of death).
Objective RR | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  Objective RR will be the best response obtained in any evaluation according to RECIST 1.1
CA-125 serological response | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  CA-125 serological response will be the best response obtained in each arm
Duration of Response | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  Duration of response: will be calculated from the date of first documentation of response (CR or partial response [PR], whichever occurs first) to the date of documented PD or death.
Time to subsequent chemotherapy administration | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  The time from randomization to subsequent chemotherapy counted from the administration of subsequent chemotherapy will be evaluated as an exploratory analysis.
OS for Subsequent chemotherapies | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  the overall survival counted from the administration of subsequent chemotherapy until death
PFS for the Subsequent Chemotherapies | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  the progression free survival counted from the administration of subsequent chemotherapy untill disease progression or death whichever occurs first
Frequency of serious adverse events (SAEs) | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  Number of SAEs for each randomization arm
QoL according to the EORTC QLQ-C30 and QLQ-OV28 | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  Two PRO instruments will be administered in this study: the EORTC QLQ-C30 and QLQ-OV28.PRO instruments will be completed by the patient at screening (before randomization) and within four weeks after the 6th cycle or at the time of progression, whichever occurs first.
Best response to each Subsequent chemotherapy line | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  The best response obtained to each Subsequent chemotherapy line calculated as frequency of patients with CR, PR, SD or PD.
Frequency of toxicities, graded according to the NCI-CTAE version 4.0 | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  Clinical and laboratory toxicities
Frequency of toxicities leading to dose delays | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  Clinical and laboratory toxicities
Frequency of toxicities leading to dose modifications | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  Clinical and laboratory toxicities
Frequency of toxicities leading to treatment discontinuation | This outcome measure will be assess approximately 4.5-5 years after the last patient enrolled, at the same time points of the Primary Endpoint
  Clinical and laboratory toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Colombo, MD, Principal Investigator — European Institute of Oncology (I.E.O), Milan, Italy
Locations (132):
- Austria (4):
  - Krankenhaus Der Barmherzigen Brueder, Graz, AT
  - Univ. Clinic for Gynaecology and Obstetrics - Medical University of Innsbruck, Innsbruck, AT
  - Medizinische Universitat Graz, Graz
  - Univ. Klinik Frauenheilkunde AKH, Vienna
- Belgium (11):
  - Imeldaziekenhuis, Bonheiden, BE
  - AZ Klina, Brasschaat, BE
  - Antwerp University Hospital, Edegem, BE
  - UZ Leuven, Leuven, BE
  - CMSE Clinique et Maternité Sainte-Elisabeth, Namur, BE
  - Az Damiaan, Ostend, BE
  - Centrum Voor Oncologie, Turnhout, BE
  - Centre Hospitalier Peltzer La Tourelle (CHPLT), Verviers, BE
  - CHU Dinant Godinne / UCL Namur, Yvoir, BE
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
- Odense University Hospital, Odense, DK, Denmark
- Finland (3):
  - Tampere University Hospital, Tampere, FI
  - Kuopio University Hospital - Kuopio, Kuopio
  - Oulu University Hospital, Oulu
- Germany (20):
  - Charite Universitaetsmedizin, Berlin, DE
  - Ev. Waldkrankenhaus Spandau, Berlin, DE
  - Praxis Dr. med. Jörg Schilling, Berlin, DE
  - Praxisklinik Krebsheilkunde für Frauen, Berlin, DE
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin, DE
  - University Hospital Dresden, Dresden, DE
  - Dr. med. Georg Heinrich Schwerpunktpraxis für Gynäkologische Onkologie, Fürstenwalde, DE
  - Kath. Marienkrankenhaus, Hamburg, DE
  - Universitäts - Frauenklinik -Tübingen, Heidelberg, DE
  - Helios Klinikum Krefeld, Krefeld, DE
  - "Universitätsklinikum Schleswig-Holstein, Lübeck, DE
  - Staedtisches Klinikum Brandenburg, Brandenburg
  - Universitatsfrauenklinik Dusseldorf, Düsseldorf
  - Kliniken Essen Mitte Evang. Huyssens Stiftung, Essen
  - University Medical Center Hamburg, Hamburg
  - Universitaetsklinikum Jena, Jena
  - Klinikum Leverkusen gGmbH, Leverkusen
  - Studienzentrum Onkologie, Ravensburg
  - UFK am Klinikum Suedstadt Rostock, Rostock
  - Onkologische Schwerpunktpraxis, Speyer
- Italy (48):
  - Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Ospedale Regionale Umberto Parini, Aosta, AO
  - "Ospedale Degli Infermi - Biella", Biella, BI
  - Policlinico S.Orsola Malpighi, Bologna, BO
  - P.O. "A.Perrino" ASL Brindisi, Brindisi, BR
  - A.O. Spedali Civili di Brescia, Brescia, BS
  - Fondazione Poliambulanza, Brescia, BS
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, CN
  - Ospedale Valduce, Como, CO
  - Azienda Ospedaliero Universitaria "Policlinico- Vittorio Emanuele" P.O. Gaspare Rodolico, Catania, CT
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) - IRCCS, Meldola e Cesena, Meldola, FC
  - Ospedale San Giuseppe - Azienda USL11, Empoli, FI
  - Ospedale SS Trinità - Sora, Sora, FR
  - Ente Ospedaliero Ospedali Galliera, Genova, GE
  - IRCCS San Martino IST - Genova, Genova, GE
  - AO della Provincia di Lecco - Ospedale Alessandro Manzoni, Lecco, LC
  - Ospedale Vito Fazzi, Lecce, LE
  - European Institute of Oncology, Department of Surgery Science, Milan, MI
  - Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, MO
  - AO Ospedali Riuniti Villa Sofia Cervello, Palermo, PA
  - Ospedale Guglielmo da Saliceto - Piacenza, Piacenza, PC
  - Istituto Oncologico Veneto, Padua, PD
  - Ospedale Santa Chiara, Pisa, PI
  - Nuovo Ospedale di Prato S. Stefano, Prato, PO
  - Istituto di Ricovero e Cura a Carattere Scientifico - Centro Regionale Oncologico Basilicata, Rionero in Vulture, PZ
  - Ospedale di Faenza, Faenza, RA
  - Ospedale Umberto I, Lugo, RA
  - Azienda Ospedaliera "Bianchi - Melacrino - Morelli", Reggio Calabria, RC
  - IRCCS - Arcispedale S. Maria Nuova, Reggio Emilia, RE
  - Policlinico Umberto I, Universitàdi Roma "La Sapienza", Roma, RM
  - Ospedale Infermi, Rimini, RN
  - Ospedale Civile di Sondrio, Sondrio, SO
  - Ospedale di Santa Chiara, Trento, TN
  - Fondazione Piemontese Per L'Oncologia - IRCCS, Candiolo, Candiolo, TO
  - AOU Città della salute e della scienza - OIRM S. Anna, Torino, TO
  - Ospedale Mauriziano, Torino, TO
  - Azienda Ospedaliero Universitaria Città Della Salute e Della Scienza di Torino - P.O. S. Anna, Torino, TO
  - Ospedale Del Ponte - Varese, Varese, VA
  - U.L.S.S. 13 Mirano - Dolo - Noale, Mirano, VE
  - Sacro Cuore Don Calabria, Negrar, VR
  - AOU Materdomini, Catanzaro
  - Università degli Studi di Napoli Federico II, Napoli
  - AOU Maggiore della Carità, Novara
  - Presidio Ospedaliero A Tortora, Pagani
  - ARNAS Civico, Palermo
  - Casa di Cura La Maddalena, Palermo
  - Ospedale S. Vincenzo, Taormina
  - ASL VC Ospedale S. Andrea - Vercelli, Vercelli
- Radboud University Medical Centre, Nijmegen, NL, Netherlands
- Norway (3):
  - Radium Hospitalet Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
- Spain (23):
  - Hospital General Universitario de Elche, Alicante, ES
  - Hospital Germans Trias I Pujol, Badalona, ES
  - Institut Català d´Oncologia, Hospitalet - Hospitalet de Llobregat, Barcelona, ES
  - Consorcio Hospitalario Provincial de Castellon, Castèllo, ES
  - Hospital Universitario Donostia - San Sebastian, Donostia / San Sebastian, ES
  - Institut Català d'Oncologia de Girona, Girona, ES
  - H. U. Arnau de Vilanova, Lleida, ES
  - MD Anderson Cancer Center, Madrid, ES
  - Althaia, Manresa, ES
  - Hospital Universitario J.M. Morales Meseguer, Murcia, ES
  - Hospital Son Espases, Palma de Mallorca, ES
  - Hospital Son Llatzer, Palma de Mallorca, ES
  - Complejo Hospitalario de Navarra, Pamplona, ES
  - Corporacion Sanitaria y Universitaria Parc Tauli, Sabadell, ES
  - Hospital General Universitario de Valencia, Valencia, ES
  - Hospital La Fe, Valencia, ES
  - IVO Instituto Valenciano de Oncologia, Valencia, ES
  - Hospital Reina Sofia, Córdoba
  - Hospital Clinico Universitario Virgen De La Arrixaca, El Palmar
  - Hospital Universitario 12 de Octubre, Madrid
  - Consorci Sanitari De Terrassa, Terrassa
  - Hospital Lluis Alcanyis Xativa, Valencia
  - Hospital Universitario Dr Peset, Valencia
- Switzerland (13):
  - Ospedale Regionale Bellinzona e Valli - Istituto Oncologico Della Svizzera Italiana (IOSI), Bellinzona, Canton Ticino
  - Kantonsspital Aarau, Aarau, CH
  - Frauenklinik -Universitätsspital Basel, Basel, CH
  - Klinik Engeried, Bern, CH
  - Universitätsklinik für Frauenheilkunde, Universitätsklinik für Onkologische Medizin - Inselspital, Bern, CH
  - Kantonsspital Graubünden, Chur, CH
  - Kantonsspital Frauenfeld, Frauenfeld, CH
  - Luzerner Kantonsspital, Lucerne, CH
  - Kantonsspital Münsterlingen, Münsterlingen, CH
  - Kantonsspital Olten, Olten, CH
  - Kantonsspital St. Gallen, Sankt Gallen, CH
  - Kantonsspital, Winterthur, CH
  - Frauenklinik - Stadtspital Triemli, Zurich, CH
- United Kingdom (5):
  - Royal Sussex County Hospital, Brighton
  - Velindre Cancer Center, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Churchill Hospital, Oxford
  - Worthingh Hospital, Worthing

REFERENCES:
- [Derived] Colombo N, Gadducci A, Sehouli J, Rulli E, Maenpaa J, Sessa C, Montes A, Ottevanger NB, Berger R, Vergote I, D'Incalci M, Churruca Galaz C, Chekerov R, Nyvang GB, Riniker S, Herbertson R, Fossati R, Barretina-Ginesta MP, Deryal M, Mirza MR, Biagioli E, Iglesias M, Funari G, Romeo M, Tasca G, Pardo B, Tognon G, Rubio-Perez MJ, DeCensi A, De Giorgi U, Zola P, Benedetti Panici P, Aglietta M, Arcangeli V, Zamagni C, Bologna A, Westermann A, Heinzelmann-Schwarz V, Tsibulak I, Wimberger P, Poveda A; INOVATYON study group. INOVATYON/ ENGOT-ov5 study: Randomized phase III international study comparing trabectedin/pegylated liposomal doxorubicin (PLD) followed by platinum at progression vs carboplatin/PLD in patients with recurrent ovarian cancer progressing within 6-12 months after last platinum line. Br J Cancer. 2023 Apr;128(8):1503-1513. doi: 10.1038/s41416-022-02108-7. Epub 2023 Feb 9. PMID 36759720